CLINICAL TRIAL: NCT05472740
Title: Transcutaneous Electrical Nerve Stimulation for Analgesia During Outpatient Endometrial Biopsy: a Randomized Controlled Trial
Brief Title: Transcutaneous Electrical Nerve Stimulation During Outpatient Endometrial Biopsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Pro00111100
Record Dates: First submitted 2022-07-22; First posted 2022-07-25 (Actual); Results first posted 2025-08-22 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Endometrial Diseases; Pain, Postoperative
Keywords: endometrial biopsy; transcutaneous electrical nerve stimulation
MeSH Terms: conditions — Uterine Diseases; Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: The participant and the provider completing the endometrial biopsy will be blinded to what group (intervention or placebo) that the subject is in. The clinical research coordinator assisting with the study and placement of the TENS will not be blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Active TENS (Experimental): Participants will be connected to a TENS 7000 that is turned on and working
  Interventions: Device: TENS 7000
- Placebo TENS (Placebo Comparator): Participants will be connected to a TENS 7000 however it will not be connected / will not be working
  Interventions: Device: TENS 7000

INTERVENTIONS:
Device: TENS 7000 — TENS device to be used in both the active and placebo groups

SUMMARY:
The purpose of this study is to see whether transcutaneous electrical nerve stimulation (or TENS) reduces pain during an endometrial biopsy. A TENS unit is an over-the-counter, FDA approved device that sends low-level electrical impulses through the skin to reduce the amount of discomfort experienced during procedures. A TENS unit is very low-risk and used in a lot of ways, including for chronic pain, after surgery, and during labor. Since there is no standard way of managing discomfort during an endometrial biopsy, the investigators think that TENS might be helpful.

Participating in the study may require some additional time in clinic to answer research-related questions. Subjects will be asked to answer demographic questions (which will be combined anonymously) before and after the procedure, as well as rate subject's pain at different time points during the procedure.

The biggest benefit in participating is that subject's discomfort might be lower during and after the procedure. Subjects may not benefit from participating in this study. There is a small risk of a skin reaction from wearing the TENS pads.

ELIGIBILITY:
Inclusion Criteria:

* at least 18 years old
* undergoing an outpatient endometrial biopsy
* Duke gynecological oncology clinics and general gynecology clinic

Exclusion Criteria:

* age younger than 18 years
* unable to follow study instructions and/or independently adjust TENS settings
* cutaneous damage at the TENS application site
* pacemaker or automatic implanted cardiac defibrillator
* inability to understand or declines to sign the informed consent form
* previous personal experience using a TENS unit
* concurrent procedure (ex. IUD placement at time of biopsy)
* pregnant women (will be excluded as part of standard of care for endometrial evaluation)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 149 (Actual)
Dates: Start 2022-12-13 (Actual); Primary Completion 2023-12-26 (Actual); Study Completion 2023-12-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Laura Havrilesky, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lerma K, Goldthwaite LM, Blumenthal PD, Shaw KA. Transcutaneous Electrical Nerve Stimulation for Pain Management of Aspiration Abortion up to 83 Days of Gestation: A Randomized Controlled Trial. Obstet Gynecol. 2021 Sep 1;138(3):417-425. doi: 10.1097/AOG.0000000000004502. PMID 34352845
- [Background] Yilmazer M, Kose S, Arioz DT, Koken G, Ozbulut O. Efficacy of transcutaneous electrical nerve stimulation for pain relief in women undergoing office endometrial biopsy. Arch Gynecol Obstet. 2012 Apr;285(4):1059-64. doi: 10.1007/s00404-011-2111-7. Epub 2011 Oct 19. PMID 22009510
- [Background] Lison JF, Amer-Cuenca JJ, Piquer-Marti S, Benavent-Caballer V, Bivia-Roig G, Marin-Buck A. Transcutaneous Nerve Stimulation for Pain Relief During Office Hysteroscopy: A Randomized Controlled Trial. Obstet Gynecol. 2017 Feb;129(2):363-370. doi: 10.1097/AOG.0000000000001842. PMID 28079781
- [Derived] Wu J, Lim S, Scott A, Hayes T, Unnithan S, Erkanli A, Havrilesky LJ, Swartz JJ. Transcutaneous Electric Nerve Stimulation for Analgesia During Outpatient Endometrial Biopsy: A Randomized Controlled Trial. Obstet Gynecol. 2025 Jan 1;145(1):e14-e23. doi: 10.1097/AOG.0000000000005727. Epub 2024 Nov 21. PMID 39575620

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Active TENS | Placebo TENS
Started | 75 | 74
Completed | 68 | 67
Not Completed | 7 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active TENS | Placebo TENS | Total
Number analyzed (Participants) | 68 | 67 | 135
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 57 | 57 | 114
  >=65 years | 11 | 10 | 21
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 68 | 67 | 135
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 16 | 26
  Not Hispanic or Latino | 58 | 51 | 109
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 5 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 34 | 23 | 57
  White | 26 | 27 | 53
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 6 | 12 | 18
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 68 | 67 | 135

OUTCOME MEASURES:

1. Primary Outcome: Pain After Endometrial Biopsy, as Measured by Visual Analogue Scale (VAS)
Description: Scores are measured on a 100 mm VAS. The VAS ranges from 0 to 100 mm with the lower score indicating less pain and the higher score indicating greater pain
Time Frame: Immediately after endometrial biopsy
Measure: Median (Inter-Quartile Range); unit: mm
Arm/Group | Active TENS | Placebo TENS
Number analyzed (Participants) | 68 | 67
mm | 50 [20 to 80] | 60 [40 to 100]
Statistical Analysis 1: Comparison: Active TENS vs Placebo TENS; Test type: Superiority; p = 0.039, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Measure of the Intervention Acceptability Based on Survey Response
Description: A 0 to 100 mm scale similar to VAS (visual analog scale) to assess acceptability of TENS (Transcutaneous Electrical Nerve Stimulation) intervention. 0 - completely acceptable to 100 - not at all acceptable
Time Frame: End of procedure
Measure: Median (Inter-Quartile Range); unit: mm
Arm/Group | Active TENS | Placebo TENS
Number analyzed (Participants) | 68 | 67
mm | 0 [0 to 22.5] | 0 [0 to 20.0]

3. Secondary Outcome: Tolerability of Procedure, as Measured by Visual Analogue Scale (VAS)
Description: A 0 to 100 mm scale similar to VAS to assess tolerability of TENS (Transcutaneous Electrical Nerve Stimulation) intervention.
Time Frame: End of procedure
Measure: Median (Inter-Quartile Range); unit: mm
Arm/Group | Active TENS | Placebo TENS
Number analyzed (Participants) | 68 | 67
mm | 17.5 [0 to 60] | 30 [0 to 70]

4. Secondary Outcome: Pain, as Measured by Visual Analogue Scale (VAS) Across Different Time Intervals
Description: as for outcome 1
Time Frame: Speculum placement, tenaculum placement, 5 minutes after biopsy, and 15 minutes after biopsy
Measure: Median (Inter-Quartile Range); unit: mm
Arm/Group | Active TENS | Placebo TENS
Number analyzed (Participants) | 68 | 67
mm
  Speculum Placement | 20 [0 to 50] | 10 [0 to 40]
  Tenaculum Placement | 50 [20 to 80] | 55 [30 to 80]
  5 min post biopsy | 10 [0 to 40] | 20 [0 to 40]
  15 min post biopsy | 7.5 [0 to 30] | 10 [0 to 30]

5. Secondary Outcome: Provider Satisfaction With the Procedure
Description: A 0 to 100 mm scale similar to VAS (visual analog scale) to assess provider satisfaction
Time Frame: End of procedure
Population: Data not collected due to unavailability of providers post-procedure.
Arm/Group | Active TENS | Placebo TENS
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse event data were collected a week after the biopsy.
Description: The study team looked for cases of post-procedural syncope, heavy bleeding, or reaction to TENS unit for a week following the biopsy. Any participant who experienced these was offered study withdrawal. Any need for hospitalization or death that was probably study related was immediately reported to the IRB.
Arm/Group | Active TENS | Placebo TENS
All-Cause Mortality (participants affected / at risk) | 0/75 | 0/74
Serious Adverse Events (participants affected / at risk) | 0/75 | 1/74
Other Adverse Events (participants affected / at risk) | 0/75 | 1/74
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active TENS (N=75) | Placebo TENS (N=74)
Esophageal dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active TENS (N=75) | Placebo TENS (N=74)
Possible electrode burn (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2023-08-23): https://cdn.clinicaltrials.gov/large-docs/40/NCT05472740/Prot_000.pdf
  • Statistical Analysis Plan (2023-08-23): https://cdn.clinicaltrials.gov/large-docs/40/NCT05472740/SAP_001.pdf
  • Informed Consent Form (2023-10-02): https://cdn.clinicaltrials.gov/large-docs/40/NCT05472740/ICF_002.pdf